CLINICAL TRIAL: NCT00128128
Title: Cranberry and Prevention of UTI A Comprehensive Approach
Brief Title: Cranberry Juice for the Prevention of Recurrent Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01AT002105-01 (NIH)
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Urinary Tract Infections
Keywords: Vaccinium macrocarpon; Cranberry; Complementary Therapies
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): Cranberry Juice Cocktail- 4 ounces
  Interventions: Drug: Cranberry juice cocktail
- Arm 2 (Active Comparator): Cranberry Juice Cocktail-8 ounces
  Interventions: Drug: Cranberry juice cocktail
- Arm 3 (Placebo Comparator): Placebo- 4 ounces
  Interventions: Drug: Cranberry juice cocktail
- Arm 4 (Placebo Comparator): Placebo- 8 ounces
  Interventions: Drug: Cranberry juice cocktail

INTERVENTIONS:
Drug: Cranberry juice cocktail — Participants will consume 4 or 8 ounces of Cranberry Juice Cocktail or Placebo daily for 6 months.
  Other Names: CJC; cranberry

SUMMARY:
This study will determine whether cranberry juice is effective in reducing recurrent urinary tract infections (UTIs) in women who have had a UTI within the past year.

DETAILED DESCRIPTION:
UTIs are a common problem among young women, resulting in considerable morbidity and health care costs. Increasing resistance to antibiotics is making treatment of these infections even more problematic. Therefore, safe and effective nonantimicrobial prevention strategies are needed. One approach that appears to be effective is the use of cranberry products. However, data on the safety and effectiveness of cranberry products are limited. This study will determine whether cranberry juice can reduce UTIs in women.

Participants will be randomly assigned to receive either cranberry juice or a placebo drink daily for 6 months. Study visits will occur every month for the 6-month treatment phase of the study. At study entry and at each study visit, urine collection will occur and vaginal swabs will be taken. A rectal swab will be taken at study entry and at the Month 2 and 4 visits. Participants will be asked about medication usage, any side effects they may be experiencing, and diet at each study visit. If participants develop a UTI at any time during the study, they will be asked to visit the study site within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* At least one UTI within 12 months prior to study entry
* Premenopausal
* Agree to avoid all foods that contain plants from the genus Vaccinium (related to cranberries) for the duration of the study

Exclusion Criteria:

* Anatomic abnormalities of the urinary tract
* History of kidney stones
* Bacteria in the urine (bacteriuria)
* Use of prophylactic antibiotics within 7 days prior to study entry
* Use of investigational drugs within 30 days prior to study entry
* Current use of warfarin
* Diabetes
* Cancer. Participants with skin cancer are not excluded.
* Allergy or intolerance of cranberry products
* Symptomatic vaginitis
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Rate of UTIs | 6 months

SECONDARY OUTCOMES:
Compliance | 6 months
vaginal and rectal colonization with E. coli | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Gupta, MD, MPH, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Stapleton AE, Dziura J, Hooton TM, Cox ME, Yarova-Yarovaya Y, Chen S, Gupta K. Recurrent urinary tract infection and urinary Escherichia coli in women ingesting cranberry juice daily: a randomized controlled trial. Mayo Clin Proc. 2012 Feb;87(2):143-50. doi: 10.1016/j.mayocp.2011.10.006. PMID 22305026
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952